CLINICAL TRIAL: NCT04554160
Title: ArrhythmiaS in Pulmonary arterIal hypeRtEnsion and Right Heart Failure Assessed by Continuous Long-term Cardiac Monitoring
Brief Title: Arrhythmias in Pulmonary Hypertension Assessed by Continuous Long-term Cardiac Monitoring
Acronym: ASPIRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Jørn Carlsen, Principal investigator, MD, DMSc, Rigshospitalet, Denmark
Other Study IDs: H-18005164
Record Dates: First submitted 2020-08-26; First posted 2020-09-18 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Hypertension; Arrhythmias, Cardiac; Heart Rate Variability; Risk Assessment
Keywords: arrhythmias; Heart rate variability; Pulmonary Hypertension; Risk assessment; Continuous heart monitoring via wearables
MeSH Terms: conditions — Hypertension, Pulmonary; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — There willl be taken 10 ml of blood for each visit (6 visits in total), of which the excess amount will be stored in a biobank. The material is stored for up to 25 years following.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Loop recorder implantation — A loop recorder is implanted in the start of the study after informed consent is signed and enables continuous cardiac monitoring.
  Other Names: Reveal LINQ loop recorder
Device: A smartwatch — A subgroup of the patients will be given an apple watch after informed consent to enables continuous monitoring via this non-invasive modality.
  Other Names: Apple watch

SUMMARY:
Arrhythmias are considered a prominent phenomenon in pulmonary hypertension (PH) as the disease progresses. According primarily to retrospective studies with up to 24 hours of monitoring, supraventricular tachycardias (SVT) can be found in 8-35% of patients, with significant impact on survival.

Furthermore, a few prospective studies to date deploying short-term monitoring (10 minutes-24 hours) have revealed lower heart rate variability (HRV) in patients with pulmonary arterial hypertension (PAH).

In ASPIRE arrhythmias and heart rate variability is being assessed via long term monitoring.

Currently the the loop-recorder is considered the gold standard for long-term continuous cardiac montoring. A non-invasive continuous monitoring could be of a great benefit for the patients, and could potentially contribute to treatment optimization.

The study will assess apple watches as a non-invasive tool compared to to the loop recorder, which is considered as the current gold standard.

Additionally, the study seeks to assess apple watches for monitoring as an independent wearable for risk assessment in PH.

DETAILED DESCRIPTION:
In general there is a lack of evidence of the arrhythmic burden in PH. The present study is the first to apply continuous long-term cardiac monitoring in patients with PH to describe the prevalence of arrhythmias in PH by continuous long-term cardiac monitoring. Furthermore, the correlation between heart rate variability and risk assessment parameters including WHO functional class (FC), NT-proBNP, 6MWT, cardiac parameters and cardiac function will be studies.

A few prospective studies have demonstrated lower HRV in PH than in healthy individuals, however only based on short-term monitoring (20 minutes to 24 hour) and only in a few patients. In retrospective studies, a higher mortality in children with PAH and low HRV has been shown with 24 hour Holter monitoring. Consequently, there is a lack of evidence regarding right heart failure and the prognostic value of HRV.

Risk assessment in PH is essential in the selection of treatment in PH and for prognosis in the study ASPIRE the investigators will assess the use of heart rate variability in pulmonary hypertension.

In conclusion the ASPIRE study will:

1. Assess the incidence and prevalence of arrhythmias using long term cardiac monitoring via a reveal LINQ loop recorder (Medtronic). Furthermore, the investigators will assess; Change in cardiac index, right atrial size, RV size, fibrosis and stroke volume.
2. The investigators will assess the arrhythmic burden in relation to:

   * Change in 6 MWT
   * Hemodynamic changes with RHC
   * Hemodynamic changes in echocardiography
   * The number of patients progressing one FC (Modified NYHA class)
   * Changes in NT-proBNP.
   * Hospital admission for any reason
   * Death or transplantation
3. Monitor heart rate variability and address a comparison to known risk markers and CMR and echocardiography.

   The study specifically seeks to investigate following:
   * The incidence and type of supraventricular and ventricular arrhythmias in PH by continuous long-term monitoring
   * The predictive value of both right and left ventricular cardiac magnetic resonance (CMR) imaging parameters for arrhythmogenesis in PAH, heart rate variability, and heart rate.
   * Optimization of specific therapy in PAH using continuous long-term arrhythmia monitoring
4. Monitor patients using smart watches (apple watches) to evaluate the applicability of long-term monitoring via apple watches in patients with pulmonary hypertension for irsk asessment.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary hypertension patients >18 years of age

  * Voluntary participation after giving informed verbal and written consent
  * Patients naïve to PAH-specific treatments
  * Patients on current PAH specific medication independent of duration of therapy
  * Patients can be in WHO group 1 classified by one of the following subgroups:
  * Idiopathic pulmonary arterial hypertension (IPAH)
  * Heritable pulmonary arterial hypertension (HPAH)
  * Drugs and toxins
  * Associated with (APAH): specifically, connective tissue disease (CTD), HIV infection and congenital heart disease
  * Patients with chronic thromboembolic pulmonary hypertension
  * Diagnosis of PAH confirmed by right heart catheterization
  * WHO/NYHA functional class II to IV symptoms
  * 6MWT distances of ≥50 meters and within 15% of each other on 2 consecutive tests preferably performed on different days during Screening.

Exclusion Criteria:

* Presence of 3 or more of the following risk factors for heart failure with preserved ejection fraction at Screening: BMI >30 kg/m2; diabetes mellitus of any type; systemic hypertension, significant coronary artery disease; or left atrial volume index (LAVi) >30 mL/m2.
* Evidence or history of left-sided heart disease and/or clinically significant cardiac disease.
* Acutely decompensated heart failure within 30 days prior to Screening
* Evidence of significant parenchymal lung disease
* Uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure (SBP) >160 mmHg or sitting diastolic blood pressure (DBP) >100 mmHg at Screening. • Systolic blood pressure >160 mmHg or < 90 mmHg; or diastolic blood pressure > 100 mgHg at Screening
* Male subjects with a corrected QT interval using Fridericia's formula (QTcF) >450 msec, and female subjects with QTcF >470 msec on ECG measured at Screening or Baseline.
* Other severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or that would confound study analysis or impair study participation or cooperation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pulmonary hypertension:
  Patients can be in WHO group 1 classified by one of the following subgroups:
  * Idiopathic pulmonary arterial hypertension (IPAH)
  * Heritable pulmonary arterial hypertension (HPAH)
  * Drugs and toxins
  * Associated with (APAH): specifically, connective tissue disease (CTD), HIV infection and congenital heart disease
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-09-24 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
The incidence and prevalence of arrhythmias in pulmonary hypertension | 2022
  Assessed throughout continuous cardiac monitoring
Heart rate variability | 2023
  Throughout continuous cardiac monitoring heart rate variability will be assessed as a clinical marker. It will be compared with already known clinical markers in pulmonary hypertension and compared with echocardiography and cardiac MR scans.
Arrhythmias and their impact on heart function assessed with echocardiography | 2022
  Change in function of the right and left heart chambers in the patients' with and without arrhythmias assessed with echocardiography.
Heart rate variability and heart function assessed with CMR scans. | 2022
  The patients' heart rate variability will be compared to the function of the right and left ventricle (LVEF, RVEF)
Heart rate variability and chamber sizes assessed CMR scans | 2023
  The patients' heart rate variability will be compared to the size of the right and left ventricle (ml)
Change in heart function when having arrhythmias, assessed with CMR scans. | 2023
  The patients' arrhythmic burden will be compared to the function of the right and left ventricle (LVEF, RVEF)
Heart size in the group with and without arrhythmias, assessed with CMR scans. | 2023
  The patients' arrhythmic burden will be compared to the size of the right and left ventricle (ml).
Chamber sizes in patients with and without arrhythmias assessed with echocardiography. | 2023
  Change in echocardiography parameters assess by the size of the right and left heart chambers (ml and cm2) in the patients with and without arrhythmias.
The association between variables recorded via the apple watch and current risk assessment parameters in PH | 2024
  Association models between the variables in order to assess the apple watch applicability for risk assessment.

SECONDARY OUTCOMES:
Arrhythmias and their impact on WHO functional class | 2022
  Modified WHO functional class when having arrhythmias

OTHER OUTCOMES:
Arrhythmias and their impact on death or transplantation | 2022
  Do any patients die because of the arrhythmias and will any patients need a transplantation because of terminal PH and arrhythmias.
Arrhythmias impact on specific PAH therapy | 2022
  How many patients will need escalation in PAH therapy when having arrhythmia and how much of an increase.
Arrhythmias impact on six minute walking tests | 2022
  Arrhythmias impact on reduction in number of meters performed in a six minute walking test during the study period.
Arrhythmias and their impact on NT-proBNP | 2022
  NT-proBNP change during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jørn Carlsen, MD, DMSC, Study Director — MD at Copenhagen University Hospital, Rigshospitalet 9- Blegdamsvej
Locations (1):
- Department of Cardiology 2141 Copenhagen University Hospital, Rigshospitalet 9- Blegdamsvej, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoeper MM, Bogaard HJ, Condliffe R, Frantz R, Khanna D, Kurzyna M, Langleben D, Manes A, Satoh T, Torres F, Wilkins MR, Badesch DB. Definitions and diagnosis of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D42-50. doi: 10.1016/j.jacc.2013.10.032. PMID 24355641
- [Background] Tongers J, Schwerdtfeger B, Klein G, Kempf T, Schaefer A, Knapp JM, Niehaus M, Korte T, Hoeper MM. Incidence and clinical relevance of supraventricular tachyarrhythmias in pulmonary hypertension. Am Heart J. 2007 Jan;153(1):127-32. doi: 10.1016/j.ahj.2006.09.008. PMID 17174650
- [Background] Wen L, Sun ML, An P, Jiang X, Sun K, Zheng L, Liu QQ, Wang L, Zhao QH, He J, Jing ZC. Frequency of supraventricular arrhythmias in patients with idiopathic pulmonary arterial hypertension. Am J Cardiol. 2014 Nov 1;114(9):1420-5. doi: 10.1016/j.amjcard.2014.07.079. Epub 2014 Aug 13. PMID 25217453
- [Background] Olsson KM, Nickel NP, Tongers J, Hoeper MM. Atrial flutter and fibrillation in patients with pulmonary hypertension. Int J Cardiol. 2013 Sep 1;167(5):2300-5. doi: 10.1016/j.ijcard.2012.06.024. Epub 2012 Jun 22. PMID 22727973
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113
- [Background] Wanamaker B, Cascino T, McLaughlin V, Oral H, Latchamsetty R, Siontis KC. Atrial Arrhythmias in Pulmonary Hypertension: Pathogenesis, Prognosis and Management. Arrhythm Electrophysiol Rev. 2018 Mar;7(1):43-48. doi: 10.15420/aer.2018.3.2. PMID 29636972
- [Background] Mercurio V, Peloquin G, Bourji KI, Diab N, Sato T, Enobun B, Housten-Harris T, Damico R, Kolb TM, Mathai SC, Tedford RJ, Tocchetti CG, Hassoun PM. Pulmonary arterial hypertension and atrial arrhythmias: incidence, risk factors, and clinical impact. Pulm Circ. 2018 Apr-Jun;8(2):2045894018769874. doi: 10.1177/2045894018769874. Epub 2018 Mar 26. PMID 29575972
- [Background] Cannillo M, Grosso Marra W, Gili S, D'Ascenzo F, Morello M, Mercante L, Mistretta E, Salera D, Zema D, Bissolino A, Fusaro E, Marra S, Libertucci D, Gaita F. Supraventricular Arrhythmias in Patients With Pulmonary Arterial Hypertension. Am J Cardiol. 2015 Dec 15;116(12):1883-9. doi: 10.1016/j.amjcard.2015.09.039. Epub 2015 Oct 9. PMID 26522342
- [Background] Cirulis MM, Ryan JJ, Archer SL. Pathophysiology, incidence, management, and consequences of cardiac arrhythmia in pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension. Pulm Circ. 2019 Jan-Mar;9(1):2045894019834890. doi: 10.1177/2045894019834890. PMID 30747032
- [Background] Rajdev A, Garan H, Biviano A. Arrhythmias in pulmonary arterial hypertension. Prog Cardiovasc Dis. 2012 Sep-Oct;55(2):180-6. doi: 10.1016/j.pcad.2012.06.002. PMID 23009914
- [Background] Folino AF, Bobbo F, Schiraldi C, Tona F, Romano S, Buja G, Bellotto F. Ventricular arrhythmias and autonomic profile in patients with primary pulmonary hypertension. Lung. 2003 Nov-Dec;181(6):321-8. doi: 10.1007/s00408-003-1034-x. PMID 14749936
- [Background] da Silva Goncalves Bos D, Van Der Bruggen CEE, Kurakula K, Sun XQ, Casali KR, Casali AG, Rol N, Szulcek R, Dos Remedios C, Guignabert C, Tu L, Dorfmuller P, Humbert M, Wijnker PJM, Kuster DWD, van der Velden J, Goumans MJ, Bogaard HJ, Vonk-Noordegraaf A, de Man FS, Handoko ML. Contribution of Impaired Parasympathetic Activity to Right Ventricular Dysfunction and Pulmonary Vascular Remodeling in Pulmonary Arterial Hypertension. Circulation. 2018 Feb 27;137(9):910-924. doi: 10.1161/CIRCULATIONAHA.117.027451. Epub 2017 Nov 22. PMID 29167228
- [Background] Lahiri MK, Kannankeril PJ, Goldberger JJ. Assessment of autonomic function in cardiovascular disease: physiological basis and prognostic implications. J Am Coll Cardiol. 2008 May 6;51(18):1725-33. doi: 10.1016/j.jacc.2008.01.038. PMID 18452777
- [Background] Vonk Noordegraaf A, Galie N. The role of the right ventricle in pulmonary arterial hypertension. Eur Respir Rev. 2011 Dec;20(122):243-53. doi: 10.1183/09059180.00006511. PMID 22130817
- [Background] Vonk-Noordegraaf A, Haddad F, Chin KM, Forfia PR, Kawut SM, Lumens J, Naeije R, Newman J, Oudiz RJ, Provencher S, Torbicki A, Voelkel NF, Hassoun PM. Right heart adaptation to pulmonary arterial hypertension: physiology and pathobiology. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D22-33. doi: 10.1016/j.jacc.2013.10.027. PMID 24355638
- [Background] Smith B, Genuardi MV, Koczo A, Zou RH, Thoma FW, Handen A, Craig E, Hogan CM, Girard T, Althouse AD, Chan SY. Atrial arrhythmias are associated with increased mortality in pulmonary arterial hypertension. Pulm Circ. 2018 Jul-Sep;8(3):2045894018790316. doi: 10.1177/2045894018790316. Epub 2018 Jul 3. PMID 29969045
- [Background] Li YH, Tholakanahalli Z, Adabag JM, Wang Z, Li J. [Effectiveness and accuracy of arrhythmia detection algorithm with the Reveal LINQ insertable cardiac monitor]. Zhonghua Xin Xue Guan Bing Za Zhi. 2018 Jun 24;46(6):470-474. doi: 10.3760/cma.j.issn.0253-3758.2018.06.011. Chinese. PMID 29925184
- [Background] Wensel R, Jilek C, Dorr M, Francis DP, Stadler H, Lange T, Blumberg F, Opitz C, Pfeifer M, Ewert R. Impaired cardiac autonomic control relates to disease severity in pulmonary hypertension. Eur Respir J. 2009 Oct;34(4):895-901. doi: 10.1183/09031936.00145708. Epub 2009 May 14. PMID 19443531
- [Background] Shaffer F, McCraty R, Zerr CL. A healthy heart is not a metronome: an integrative review of the heart's anatomy and heart rate variability. Front Psychol. 2014 Sep 30;5:1040. doi: 10.3389/fpsyg.2014.01040. eCollection 2014. PMID 25324790
- [Background] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Background] Smilde TD, van Veldhuisen DJ, van den Berg MP. Prognostic value of heart rate variability and ventricular arrhythmias during 13-year follow-up in patients with mild to moderate heart failure. Clin Res Cardiol. 2009 Apr;98(4):233-9. doi: 10.1007/s00392-009-0747-0. Epub 2009 Feb 13. PMID 19219394
- [Background] Huikuri HV, Stein PK. Heart rate variability in risk stratification of cardiac patients. Prog Cardiovasc Dis. 2013 Sep-Oct;56(2):153-9. doi: 10.1016/j.pcad.2013.07.003. Epub 2013 Aug 12. PMID 24215747
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Galinier M, Pathak A, Fourcade J, Androdias C, Curnier D, Varnous S, Boveda S, Massabuau P, Fauvel M, Senard JM, Bounhoure JP. Depressed low frequency power of heart rate variability as an independent predictor of sudden death in chronic heart failure. Eur Heart J. 2000 Mar;21(6):475-82. doi: 10.1053/euhj.1999.1875. PMID 10681488
- [Background] Lammers AE, Munnery E, Hislop AA, Haworth SG. Heart rate variability predicts outcome in children with pulmonary arterial hypertension. Int J Cardiol. 2010 Jul 9;142(2):159-65. doi: 10.1016/j.ijcard.2008.12.087. Epub 2009 Jan 26. PMID 19176261
- [Background] Umetani K, Singer DH, McCraty R, Atkinson M. Twenty-four hour time domain heart rate variability and heart rate: relations to age and gender over nine decades. J Am Coll Cardiol. 1998 Mar 1;31(3):593-601. doi: 10.1016/s0735-1097(97)00554-8. PMID 9502641
- [Background] Florea VG, Cohn JN. The autonomic nervous system and heart failure. Circ Res. 2014 May 23;114(11):1815-26. doi: 10.1161/CIRCRESAHA.114.302589. PMID 24855204
- [Background] Jankowska EA, Ponikowski P, Piepoli MF, Banasiak W, Anker SD, Poole-Wilson PA. Autonomic imbalance and immune activation in chronic heart failure - pathophysiological links. Cardiovasc Res. 2006 Jun 1;70(3):434-45. doi: 10.1016/j.cardiores.2006.01.013. Epub 2006 Feb 14. PMID 16480965
- [Background] Yi HT, Hsieh YC, Wu TJ, Huang JL, Lin WW, Liang KW, Su CS, Tsai WJ, Wang KY. Heart rate variability parameters and ventricular arrhythmia correlate with pulmonary arterial pressure in adult patients with idiopathic pulmonary arterial hypertension. Heart Lung. 2014 Nov-Dec;43(6):534-40. doi: 10.1016/j.hrtlng.2014.05.010. Epub 2014 Jun 11. PMID 24929769
- [Background] Fauchier L, Babuty D, Melin A, Bonnet P, Cosnay P, Paul Fauchier J. Heart rate variability in severe right or left heart failure: the role of pulmonary hypertension and resistances. Eur J Heart Fail. 2004 Mar 1;6(2):181-5. doi: 10.1016/j.ejheart.2003.09.007. PMID 14984725
- [Background] Tsai CH, Ma HP, Lin YT, Hung CS, Hsieh MC, Chang TY, Kuo PH, Lin C, Lo MT, Hsu HH, Peng CK, Lin YH. Heart Rhythm Complexity Impairment in Patients with Pulmonary Hypertension. Sci Rep. 2019 Jul 24;9(1):10710. doi: 10.1038/s41598-019-47144-1. PMID 31341216
- [Background] Weatherald J, Boucly A, Sitbon O. Risk stratification in pulmonary arterial hypertension. Curr Opin Pulm Med. 2018 Sep;24(5):407-415. doi: 10.1097/MCP.0000000000000510. PMID 30004992
- [Background] Chin KM, Rubin LJ, Channick R, Di Scala L, Gaine S, Galie N, Ghofrani HA, Hoeper MM, Lang IM, McLaughlin VV, Preiss R, Simonneau G, Sitbon O, Tapson VF. Association of N-Terminal Pro Brain Natriuretic Peptide and Long-Term Outcome in Patients With Pulmonary Arterial Hypertension. Circulation. 2019 May 21;139(21):2440-2450. doi: 10.1161/CIRCULATIONAHA.118.039360. PMID 30982349
- [Background] Sanders P, Purerfellner H, Pokushalov E, Sarkar S, Di Bacco M, Maus B, Dekker LR; Reveal LINQ Usability Investigators. Performance of a new atrial fibrillation detection algorithm in a miniaturized insertable cardiac monitor: Results from the Reveal LINQ Usability Study. Heart Rhythm. 2016 Jul;13(7):1425-30. doi: 10.1016/j.hrthm.2016.03.005. Epub 2016 Mar 4. PMID 26961298
- [Background] Andrade J, Khairy P, Dobrev D, Nattel S. The clinical profile and pathophysiology of atrial fibrillation: relationships among clinical features, epidemiology, and mechanisms. Circ Res. 2014 Apr 25;114(9):1453-68. doi: 10.1161/CIRCRESAHA.114.303211. PMID 24763464

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT04554160/Prot_SAP_000.pdf